CLINICAL TRIAL: NCT02933359
Title: Osteogenic Profiling of Normal Calvarial Bone
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Joseph Losee, Professor of Surgery, University of Pittsburgh
Other Study IDs: PRO10070450
Record Dates: First submitted 2016-08-22; First posted 2016-10-14 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Fracture; Skull
Keywords: cranial vault; calvarial trauma; calvarial reconstruction
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone samples will be collected from bone tissue that would normally be discarded during the reconstructive surgery, so no additional procedures are needed to collect the bone samples. Bone marrow tissues will be collected from patients at the time of surgery without any additional dissection or incisions. Bone will be finely minced and then plated in tissue culture flasks as previously reported by other groups.
  The procedure will not involve any extra incisions or dissection, as these tissues will be exposed during the reconstructive procedure. At the time of surgery one sample of tissue will be taken from otherwise discarded bone
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal Tissue: Bone fragments and their associated bone marrow will be collected from patients at the time of surgery without any additional dissection or incisions. Bone will be finely minced and then plated in tissue culture flasks as previously reported by other groups [7].

SUMMARY:
The primary objectives of this study are:

i) to procure human calvarial bone, ii) to grow cells from these tissues in vitro, iii) and to evaluate the osteogenic potential of these cells.

DETAILED DESCRIPTION:
For outpatient study recruitment, the research coordinator will review the clinic schedule for potential study candidates. Any patient schedule for a pre-op appointment for surgical calvarial reconstruction will be considered a possible study candidate. The research coordinator will then e-mail the study team the list of potential study candidates with the date and time of the appointment or in-patient study recruitment, the screening procedures include review and collection of information from the patient's medical record-specifically, a physical examination by the plastic surgeon at the Cleft Palate-Craniofacial Center Plastic surgery department. This evaluation will occur either as an inpatient or as an outpatient, depending on the appropriateness and timing of the ultimate surgical repair. During the clinical examination, the plastic surgeon will determine if portions of the skull are unusable for reconstruction. These bone fragments (when too small or shattered to be incorporated into a reconstruction) are normally discarded. It is these fragments alone that will be harvested for evaluation in the present study. The evaluation and surgical repair of these patients requiring post-traumatic reconstruction will not differ from normal, nor from the current standard of care.

Bone samples will be collected from bone tissue that would normally be discarded during the reconstructive surgery, so no additional procedures are needed to collect the bone samples. At the time of surgery one sample of tissue will be taken from bone. The investigator will review the results of the test/procedure that are part of the standard of care and results will become part of the research record. The investigators will continue to use and disclose identifiable medical information and keep tissue samples for seven years. After this seven year period, all identifying information will be removed. Bone marrow tissues will be collected from patients at the time of surgery without any additional dissection or incisions. Bone will be finely minced and then plated in tissue culture flasks as previously reported by other groups.

The procedure will not involve any extra incisions or dissection, as these tissues will be exposed during the reconstructive procedure. At the time of surgery one sample of tissue will be taken from otherwise discarded bone.

Samples will be collected and coded by the plastic surgeon/principal investigator before transfer from the operative room to the Pediatric Craniofacial Biology Laboratory.

The research coordinator will notify Dr. Bykowski of when consented subjects are scheduled for surgery via e-mail. Dr. Bykowski will collect the coded sample and transport them to the Pediatric Craniofacial Biology laboratory.

Cells from each tissue sample will be cultured in vitro. These cells will eventually be kept and frozen in this lab in a temperature locked freezer. The Research Assistant Professor will record subject information into a secure database in Pediatric Craniofacial Biology Laboratory. No information permitting personal identification of family members will be made public. No clinical descriptions that might permit personal identifications will be published, and all clinical information will be stored in secure computer files in the Pediatric Craniofacial Biology Laboratory, which are password protected. Specimens will be stored with assigned code numbers and information linking theses code numbers to the corresponding subjects' identities will also be kept in a password protected database. If a subject should decide to withdraw or be withdrawn from study participation, the linkage code to subject's identity and the specimen will be destroyed.

All cells will be grown in one of two media. Proliferation medium will be used during cell isolation and expansion and will consist of Dulbecco's Modified Eagle's Medium (DMEM) supplemented with 10% fetal bovine serum (FBS), and 1% penicillin/streptomycin. For mineralization studies, cells will be grown in osteogenic medium (OM) consisting of DMEM supplemented with 10% FBS, 1% penicillin/streptomycin, 10mM β-glycerophosphate, 0.1μM dexamethasone, 50μg/ml ascorbic acid-2-phosphate.

Solid-phase printed arrays of square-shaped 'blots' of immobilized BMP2 will be printed on sialanized fibrin-coated glass cover slips. The blots will be 750 um x 750 um and spaced 1.75 mm apart in a 4 x 4 array. There will be blots with 4 different concentrations of BMP2, ranging from zero to binding site saturation, along each column, and there will be 4 replicates of each column.

The homogenous fibrin films cross-linked to glass slides will be prepared. Blot concentrations will be modulated using the overprinting strategy. Pattern accuracy and surface concentration of growth factors and their persistence will be verified for FGF2. BMP2 bio-inks will be diluted to 10 µg/ml in 20 mM sodium acetate, pH 7.4. Preliminary experiments on immobilization and persistence of BMP2 on fibrin films indicate at least 6 day persistence.

Bio-ink Formulations for BMP2 and Inhibitors. The purpose here is to determine the concentration and to provide initial validation of patterned inhibition response. FGF2 bio-inks will be prepared. All bio-inks will be diluted to a 10 µg/ml. Since the number of binding sites on a square is fixed, the bio-ink dilutions and/or number of overprints may be modified based on initial results to accommodate multiple growth factors now occupying a given square. From the above array studies the investigators will determine the concentrations of BMP2 and inhibitor necessary to show stimulation/inhibition.

Cells will be placed on the printed patterns described above. Cells grown on discreet arrays will be fixed and stained for ALP activity (Sigma) after 1, 3, or 7 days in culture on the growth factor patterns. Mineralization will be tested after culturing cells on patterns in OM for 7, 14, or 21 days using alizarin red staining (for calcium) and von Kossa staining (for phosphates). ALP staining will be performed to identify early osteogenic differentiation. To signify "end" of BMP2 signaling, matrix mineralization will be determined by positive von Kossa or alizarin red staining using established protocols.

BMP2 and potential inhibitor proteins can be deposited simultaneously. The image pattern for jetting the array will be the same as in Figures 1 and 3, with the image pattern for the inhibitor being the same as the BMP2 pattern, only rotated by 90°. The jetting will be coordinated with the stage motions so that these two patterns will exactly overlap using computer-vision calibration. Pattern accuracies will be verified using fluorescently-labeled BMP2 and inhibitors.

The concentrations of BMP2 that are capable of inducing ALP activity and matrix mineralization and the concentrations of inhibitors that are capable of counteracting BMP2-induced osteogenesis will be identified and recorded for each patient. In comparing the respective osteogenic potentials, the investigators will develop "osteogenic profiles" for each of the tissue samples isolated from the patients

ELIGIBILITY:
Inclusion Criteria:

* All patients between the ages of 2 months of age to 18 years with the diagnosis of pre-operative calvarial defect secondary to trauma and undergoing surgical calvarial reconstruction will be asked to contribute to this study.

Exclusion Criteria:

* All patient with a concurrent diagnosis of craniosynostosis or other craniofacial anomaly and any child with calvarial trauma that is not undergoing surgical calvarial reconstruction will be excluded from this study

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with calvarial trauma (an insult which disrupts the cranial vault requiring surgical management to correct the injury) undergoing surgical calvarial reconstruction between the ages of 2 months of age to 18 years old will be included in this study. Children will be evaluated initially at the Pittsburgh Cleft Palate and Craniofacial Center at Children's Hospital of Pittsburgh which is set up to accommodate children of all ages and their families.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Cell Growth | 2 years
  to grow cells from the calvarial bone in vitro and freeze these collected cells for DNA analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Pittsburgh Of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data

REFERENCES:
- [Background] Whitaker LA, Munro IR, Salyer KE, Jackson IT, Ortiz-Monasterio F, Marchac D. Combined report of problems and complications in 793 craniofacial operations. Plast Reconstr Surg. 1979 Aug;64(2):198-203. doi: 10.1097/00006534-197908000-00011. PMID 377338
- [Result] Thorne, C., Grabb, W.C., and Smith, J.W. 2007. Grabb and Smith's plastic surgery. Philadelphia: Wolters Kluwer Health/Lippincott Williams & Wilkins.
- [Result] Crysdale WS, Kohli-Dang N, Mullins GC, Pullerits J, Munro IR, Burke RC. Airway management in craniofacial surgery: experience in 542 patients. J Otolaryngol. 1987 Aug;16(4):207-15. PMID 3656500
- [Result] Prevot M, Renier D, Marchac D. Lack of ossification after cranioplasty for craniosynostosis: a review of relevant factors in 592 consecutive patients. J Craniofac Surg. 1993 Oct;4(4):247-54; discussion 255-6. PMID 8110906
- [Result] Dudas JR, Marra KG, Cooper GM, Penascino VM, Mooney MP, Jiang S, Rubin JP, Losee JE. The osteogenic potential of adipose-derived stem cells for the repair of rabbit calvarial defects. Ann Plast Surg. 2006 May;56(5):543-8. doi: 10.1097/01.sap.0000210629.17727.bd. PMID 16641633
- [Result] Zuk PA, Zhu M, Mizuno H, Huang J, Futrell JW, Katz AJ, Benhaim P, Lorenz HP, Hedrick MH. Multilineage cells from human adipose tissue: implications for cell-based therapies. Tissue Eng. 2001 Apr;7(2):211-28. doi: 10.1089/107632701300062859. PMID 11304456
- [Result] Petrie C, Tholpady S, Ogle R, Botchwey E. Proliferative capacity and osteogenic potential of novel dura mater stem cells on poly-lactic-co-glycolic acid. J Biomed Mater Res A. 2008 Apr;85(1):61-71. doi: 10.1002/jbm.a.31367. PMID 17688255
- [Result] Campbell PG, Miller ED, Fisher GW, Walker LM, Weiss LE. Engineered spatial patterns of FGF-2 immobilized on fibrin direct cell organization. Biomaterials. 2005 Nov;26(33):6762-70. doi: 10.1016/j.biomaterials.2005.04.032. PMID 15941581
- [Result] Miller ED, Fisher GW, Weiss LE, Walker LM, Campbell PG. Dose-dependent cell growth in response to concentration modulated patterns of FGF-2 printed on fibrin. Biomaterials. 2006 Apr;27(10):2213-21. doi: 10.1016/j.biomaterials.2005.10.021. Epub 2005 Dec 1. PMID 16325254
- [Result] Jadlowiec J, Koch H, Zhang X, Campbell PG, Seyedain M, Sfeir C. Phosphophoryn regulates the gene expression and differentiation of NIH3T3, MC3T3-E1, and human mesenchymal stem cells via the integrin/MAPK signaling pathway. J Biol Chem. 2004 Dec 17;279(51):53323-30. doi: 10.1074/jbc.M404934200. Epub 2004 Sep 13. PMID 15371433
- [Result] Higuchi C, Myoui A, Hashimoto N, Kuriyama K, Yoshioka K, Yoshikawa H, Itoh K. Continuous inhibition of MAPK signaling promotes the early osteoblastic differentiation and mineralization of the extracellular matrix. J Bone Miner Res. 2002 Oct;17(10):1785-94. doi: 10.1359/jbmr.2002.17.10.1785. PMID 12369782